CLINICAL TRIAL: NCT02680470
Title: Virtual Observed Therapy for Patients With Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15/WS/0004
Record Dates: First submitted 2016-01-28; First posted 2016-02-11 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Management; Observed therapy
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual Observed Therapy (Experimental): Intervention = Virtual observed therapy of participants taking TB therapy
  Interventions: Device: Virtual observed therapy

INTERVENTIONS:
Device: Virtual observed therapy — Virtual Observation of participants taking their medication

SUMMARY:
Using modern technology, investigators will observe participants taking their TB tablets three times per week using a mobile phone, iPod or computer with camera facilities in the participants home environment.

DETAILED DESCRIPTION:
Using modern technology, the investigators will observe participants taking their TB tablets three times per week using a mobile phone, iPod or computer with camera facilities in the participants home environment.

Investigators will connect to the participants mobile phone, iPod or computer at a mutually convenient time three times per week who will observe participants taking their TB medication.

The Virtual Observed Therapy will be carried out using NHS Lothian approved software (mobile app called POLYCOM) three times per week. This is software similar to Skype but POLYCOM is the approved software we use in NHS Lothian.

ELIGIBILITY:
Inclusion Criteria:

Any patient requiring Tuberculosis treatment

Exclusion Criteria:

Those refusing consent; the healthcare professional deems the patient that will not be able to comply with VOT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Treatment completion rates using VOT compared with historical completion rates. | length of TB treatment (usually 6-12 months)

SECONDARY OUTCOMES:
% Cure from TB treatment | length of TB treatment (usually 6-12 months)
number of VOT actually observed divided by the expected VOT observed | length of TB treatment (usually 6-12 months)
patient satisfaction questionnaire at end of treatment | length of TB treatment (usually 6-12 months)
Mortality | length of TB treatment (usually 6-12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No